CLINICAL TRIAL: NCT03792334
Title: A Comparison Between Patient State Index (PSI) and Bispectral Index (BIS) as Technologies for Monitor in Depth of Anesthesia in Children: A Prospective Observational Trial
Brief Title: Comparison of BIS and PIS in Children
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Soo Kim, Principal Investigator, Seoul National University Hospital
Other Study IDs: 1811-172-991
Record Dates: First submitted 2018-12-28; First posted 2019-01-03 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2019-01

CONDITIONS: Depth of Anesthesia Monitor

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: depth of anesthesia — monitoring of depth of anesthesia

SUMMARY:
Comparison of bispectral index and patient sedation index during general anesthesia in children

DETAILED DESCRIPTION:
the values of BIS and PSI of every 1 minute during general anesthesia in children

ELIGIBILITY:
Inclusion Criteria:

* general anesthesia

Exclusion Criteria:

* developmental delay
* IICP

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: general anesthesia
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2019-12-26 (Actual); Study Completion 2019-12-28 (Actual)

PRIMARY OUTCOMES:
correlation of BIS and PSI | through study completion, an average of 2 hours
  difference of BIS and PSI values

CONTACTS AND LOCATIONS:
Overall Officials: Hee-Soo Kim, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (2):
- South Korea (2):
  - SNUH, Seoul, Jongnogu
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jang YE, Kim EH, Lee JH, Kim JT, Kim HS. Usefulness of bispectral index and patient state index during sevoflurane anesthesia in children: A prospective observational study. Medicine (Baltimore). 2022 Jul 29;101(30):e29925. doi: 10.1097/MD.0000000000029925. PMID 35905224